CLINICAL TRIAL: NCT06582979
Title: The Effect of Combined Intervention (Indonesian Computer-Based Game Therapy and High-Intensity Interval Training) Towards Clinical Symptoms, Executive Function and Neuroplasticity in Adolescents with Internet Gaming Disorder: Study Protocol
Brief Title: Effect of Computer-Based Game and HIIT Towards Symptoms, Executive Function and Neuroplasticity in Teens with IGD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, A M Y Eva Suryani, Eva Suryani, dr., Sp.KJ, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-03-0436
Record Dates: First submitted 2024-08-31; First posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Internet Gaming Disorder
Keywords: Indonesia; Computer-based game; High-Intensity Interval Training; Executive Function; Neuroplasticity; Adolescents; Internet Gaming Disorder; Study protocol; Teens
MeSH Terms: conditions — Internet Addiction Disorder | interventions — High-Intensity Interval Training

STUDY DESIGN:
Intervention Model Description: One group pre and post-test design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined Intervention Group (Experimental): This group will experience both computer-based game therapy and also high-intensity interval training for 7 weeks.
  Interventions: Behavioral: Computer-Based Game Therapy; Behavioral: High-Intensity Interval Training

INTERVENTIONS:
Behavioral: Computer-Based Game Therapy — Computer-based game intervention will be done three times a week, every morning before school lessons begin or during break time. Researchers will give a brief explanation of the rules on how to play the game before the intervention begins. In the game, participants will act as a fruit truck delivery driver and will have to sort out fruit delivery to different houses according to the instructions of the game. For example, the instruction starts with delivering a yellow-colored banana to a house with a red-colored roof, or delivering a purple-colored grape to a house with a blue-colored roof. Participants will first have to finish a minimum of three tutorial rounds reaching ≥75% correct delivery. Instructions will be divided into four stages; visual stimulus, auditory stimulus, visual stimulus with an obstacle, auditory stimulus with an obstacle. Each round will last for 2 minutes. Total time needed to complete a single computer-based intervention session is around 30-45 minutes.
Behavioral: High-Intensity Interval Training — HIIT will be done two times a week during physical education hours (in the school's sports field) led by the school's physical education teacher and also certified physical trainers who have undergone training supervised by a sports medicine physician. Before the start of each HIIT session, participants will have their pulse rate assessed with a pulse oximetry and then undergo warm-up for 5 minutes. The duration of each HIIT session will be continuously extended starting at around 4 minutes (1 tabata block/8 moves) during the first week to 8 minutes (2 tabata block/16 moves) during the final week. A single tabata block moveset incorporates 8 total moves; squat jump, push up, high skipping, burpees, isometric front plank, multi jumps on bench, mountain climber in hand plank and lateral sprint (5m). Each move will be done for 20 seconds, followed by a 10 second rest. Pulse rate will be assessed again after the HIIT session and then participants will undergo cooling down and relaxation.

SUMMARY:
The goal of this clinical trial is to learn how effective a combined therapy of computer-based game and also high-intensity interval training (HIIT) physical exercise to improve the clinical symptoms, executive function and neuroplasticity in teenagers with Internet Gaming Disorder (IGD). Executive function refers to the brain's ability to manage tasks such as planning, problem-solving, and decision-making. BDNF is a protein crucial for brain health and development. Neuroplasticity is the brain's ability to change and adapt throughout life. High-intensity interval training involves short bursts of intense exercise followed by periods of rest or recovery. The main questions it aims to answer are:

* How effective are computer-based game and HIIT exercises in reducing addiction symptoms of IGD?
* Will computer-based game and HIIT exercise help teens who are addicted to video games to improve their executive function (become more able to plan ahead and meet goals, display self-control and also follow multiple-step directions)?
* Do computer-based game and HIIT exercise help brains of teens with IGD to be more able to change and adapt?

Researchers will compare the improvement before and after the therapies.

Participants will:

* Undergo both therapies (computer-based game and HIIT) every week for 7 weeks. Computer-based game will be done 3 times/week and HIIT 2 times/week
* fill out forms, interviewed and also have their blood sample taken for a total of three times (before the start of the therapy, during the 4th week of therapy and after the final therapy session on the 7th week)

DETAILED DESCRIPTION:
This is a study protocol of a clinical study to examine the effectiveness of computer-based game and high-intensity interval training towards improvement of clinical symptoms, executive function and neuroplasticity in adolescents with Internet Gaming Disorder (IGD).

According to calculations, our study will aim for a minimum of 44 participants using purposive sampling. Participants will drop-out of the study if they missed >10% participation (>3 sessions out of 35 total sessions). Analysis of the effectiveness of both interventions (computer-based game and HIIT exercise) on improvement of clinical symptoms of Internet Gaming Disorder will be done using McNemar test. Meanwhile, analysis of the effectiveness of both interventions towards executive function and neuroplasticity will be done using paired-T tests. Significance levels will be set at 0.05 for analysis. All data will be analyzed using IBM SPSS v. 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Participants who have filled and agreed to the study by signing the informed assent.
* Parents of the participants have filled and agreed to the interventions by signing the informed consent.
* Participants able to follow instruction and procedure of the study

Exclusion Criteria:

* Physical disabilities
* Hearing disabilities
* Color blindness
* Respiratory or cardiovascular comorbidities that hinders exercise abilities
* Other psychiatric comorbidities

Ages: 13 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2025-01-16 (Estimated); Primary Completion 2025-03-06 (Estimated); Study Completion 2025-07-21 (Estimated)

PRIMARY OUTCOMES:
Clinical Symptoms | Baseline (T0), 4th week of intervention (T1), 7th week of intervention (T2)
  Clinical Symptoms of Internet Gaming Disorder evaluated with Ten-Item Internet Gaming Disorder Test (IGDT-10) questionnaire
Executive Function | Baseline (T0), 4th week of intervention (T1), 7th week of intervention (T2)
  Executive Function assessed with Behavior Rating Inventory of Executive Function (BRIEF) questionnaire
Neuroplasticity | Baseline (T0), 4th week of intervention (T1), 7th week of intervention (T2)
  Neuroplasticity measured with serum brain-derived neurotrophic factor (BDNF) levels

CONTACTS AND LOCATIONS:
Overall Officials: Eva Suryani, dr., Sp.KJ., Principal Investigator — Doctoral Program, Faculty of Medicine, Universitas Indonesia/Dr. Cipto Mangunkusumo General Hospital
Locations (1):
- Faculty of Medicine, Universitas Indonesia - Dr. Cipto Mangunkusumo General Hospital, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No